CLINICAL TRIAL: NCT01300130
Title: Investigations on Improving Docosahexaenoic and Arachidonic Acid Content in Preterm Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry); German Federal Ministry of Education and Research (Other Government); German Research Foundation (Other)
Responsible Party: Ludwig-Maximilians - University of Munich, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 45-95
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Prematurity of Fetus
Keywords: neurological development; preterm infants; fatty acid status
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- low docosahexaenoic acid formula (Experimental)
  Interventions: Dietary Supplement: low docosahexaenoic acid formula
- medium docosahexaenoic acid formula (Experimental)
  Interventions: Dietary Supplement: medium docosahexaenoic acid formula
- high docosahexaenoic acid formula (Experimental)
  Interventions: Dietary Supplement: high docosahexaenoic acid formula
- human milk (Active Comparator)
  Interventions: Dietary Supplement: breast milk

INTERVENTIONS:
Dietary Supplement: low docosahexaenoic acid formula
  Arms: low docosahexaenoic acid formula
Dietary Supplement: medium docosahexaenoic acid formula
  Arms: medium docosahexaenoic acid formula
Dietary Supplement: high docosahexaenoic acid formula
  Arms: high docosahexaenoic acid formula
Dietary Supplement: breast milk — a non randomized group of breast milk fed infants was included
  Arms: human milk

SUMMARY:
The investigators examined the effect of different levels of docosahexaenoic aicd (a long chain polyunsaturated fatty acid) intake on the fatty acid composition of plasma and erythrocyte phospholipids and on the maturity of visually evoked potentials in preterm infants. As a secondary outcome the conversion of linoleic acid and alpha linolenic acid into their corresponding long chain polyunsaturated fatty acids was studied.

Preterm infants were randomized in a double-blind fashion to one of three formulas containing different amounts of docosahexaenoic acid during the first two weeks of postnatal life. A control group received human milk. Blood samples were collected at study entry and 14 and 28 days thereafter. Uniformly 13C-labeled linoleic acid and alpha linolenic acid were applied orally before blood sampling at day 28. At postconceptional ages 48 weeks and 56 weeks visually evoked potentials were recorded.

ELIGIBILITY:
Inclusion Criteria:

* preterm birth
* birth weight between 1000 and 2200 g
* more than 80 % of energy intake from infant formula or human milk at enrollment

Exclusion Criteria:

* apparent genetic, gastrointestinal or metabolic disorders
* artificial ventilation or oxygen supply > 30% at the time of enrollment
* administration of parenteral fat emulsion (> 1 g/kg/day for more than seven days) before or after study entry

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 1995-06; Primary Completion 1998-03 (Actual); Study Completion 1998-03 (Actual)

PRIMARY OUTCOMES:
plasma phospholipid fatty acid composition | 28 days after intervention start
visually evoked potentials | 48 weeks and 56 weeks postconceptional age

SECONDARY OUTCOMES:
intensity of endogenous conversion of essential fatty acids into long chain polyunsaturated fatty acids | 28 days after study start

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (5):
- Germany (5):
  - Children´s Hospital, Zentralklinikum Augsburg, Augsburg
  - Josephinum Hospital, Augsburg
  - I. Frauenklinik of the Ludwig-Maximilians-University, München
  - Lachnerklinik, München
  - University Hospital Rechts der Isar, München

REFERENCES:
- [Derived] Sauerwald UC, Fink MM, Demmelmair H, Schoenaich PV, Rauh-Pfeiffer AA, Koletzko B. Effect of different levels of docosahexaenoic acid supply on fatty acid status and linoleic and alpha-linolenic acid conversion in preterm infants. J Pediatr Gastroenterol Nutr. 2012 Mar;54(3):353-63. doi: 10.1097/MPG.0b013e31823c3bfd. PMID 22008957